CLINICAL TRIAL: NCT05419830
Title: Sleep, Hypertension, and Nocturia: a Multicomponent Approach for Comorbid Illnesses
Acronym: SHyN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shachi Tyagi, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY21050132; 1R33AG057806 (NIH)
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Nocturia; Hypertension; Sleep Disturbance
MeSH Terms: conditions — Nocturia; Hypertension; Parasomnias | interventions — Chronotherapy

STUDY DESIGN:
Intervention Model Description: In the proposed pilot study 30 community-dwelling older adults (aged >65) who take at ≥1 daily non-diuretic antihypertensive medication, have a mean SBP >135 mm Hg, and awaken ≥2 times nightly to void will be randomly assigned to one of the 3 groups of 10 participants each to 1) morning (am) HTN medication dosing, 2) BBTI with am HTN medication dosing, 3) nighttime non-diuretic HTN medication dosing (chronotherapy) for 6 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization envelopes will be prepared by the study statistician. Randomization and the intervention BBTI will be completed by research nurse and PI and the outcome assessor will be blinded to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AM (morning) antihypertensive dosing arm or Control arm (Active Comparator): participants will be asked to continue taking their antihypertensive medication within an hour of awakening
  Interventions: Other: AM antihypertensive dosing
- BBTI arm (Experimental): participants will receive the behavioral treatment for insomnia BBTI by the study nurse. Participants will also be asked to take their antihypertensive medication within an hour of awakening
  Interventions: Behavioral: BBTI
- PM (evening) antihypertensive dosing or Chronotherapy arm (Experimental): participants will be asked to switch their conventional once daily non-diuretic antihypertensive to bedtime
  Interventions: Other: PM antihypertensive dosing or Chronotherapy

INTERVENTIONS:
Behavioral: BBTI — Participants randomized to BBTI will receive 45- to 60-minute individual intervention session followed by a 30-minute follow-up session 2 weeks later, and 20-minute telephone calls after 1 and 3 weeks. BBTI will focus on four behaviors that promote sleep and discussion of homeostatic and circadian mechanisms of human sleep regulation. These four interventions are simple to conceptualize and implement, and constitute the core of efficacious multi-modal behavioral treatments for insomnia.
  Arms: BBTI arm
Other: PM antihypertensive dosing or Chronotherapy — participants will be asked to switch their conventional once daily non-diuretic antihypertensive to bedtime
  Arms: PM (evening) antihypertensive dosing or Chronotherapy arm
Other: AM antihypertensive dosing — participants will be asked to continue taking their antihypertensive medication within an hour of awakening
  Arms: AM (morning) antihypertensive dosing arm or Control arm

SUMMARY:
In this study the investigators target three common and comorbid illnesses among older adults namely nocturia or waking at night to void, poor sleep and hypertension. The aim of this proposal is to test behavioral sleep intervention to improve sleep and nocturia vs switching the time of antihypertensive administration to improve nighttime and in turn daytime blood pressure control.

DETAILED DESCRIPTION:
The investigators posit that a vicious cycle operates between nocturia, poor sleep, and nighttime hypertension (HTN). HTN act through the pressure-natriuresis mechanism that links sodium (Na) and BP homeostasis: periodic increases in BP drive compensatory renal excretion of Na (natriuresis) and water (diuresis) to reduce blood volume and BP. Normally, BP and natriuresis declines during sleep, decreasing nighttime urine volume (NUV). Elevated nighttime BP increases nocturnal natriuresis causing an increase in nighttime urine volume and hence, NP: the major etiologic factor for nocturia in the elderly. In a recently completed study (AG050892, PI:Tyagi), it was found that poor sleep blunts the normal nighttime rise in antidiuretic hormone-a potent Na conserving hormone, which leads to nocturnal natriuresis and, as a result, NP. Hence, our model incorporates the effects of poor sleep and nighttime HTN on natriuresis, NP, and nocturia. The investigators postulate that treatments targeted towards these etiologies will help break this vicious cycle.

Traditionally, antihypertensive medications are dosed in the morning targeting daytime BP. However, some research suggests that nighttime BP best predicts risk for major cardiovascular events. Several clinical trials of bedtime dosing of BP medication-chronotherapy- show better nighttime BP control. However, no clinical studies have considered or tested chronotherapy as a treatment for nocturia. With respect to poor sleep, the investigators have shown that brief behavioral treatment of insomnia (BBTI) significantly improves not only sleep but also self-reported nocturia among the elderly. Therefore, the investigators envision a multicomponent approach with chronotherapy (bedtime dosing of certain antihypertensives) and behavioral sleep intervention (BBTI) to concurrently address the prevalent and chronic, mutually exacerbating conditions: nocturia, poor sleep, and HTN. The current proposal aims to collect pilot data for a definitive randomized clinical trial.

In the proposed pilot study 30 community-dwelling older adults (aged >65) who take at ≥1 daily non-diuretic antihypertensive medication, have a mean SBP >135 mm Hg, and awaken ≥2 times nightly to void will be randomly assigned to one of the 3 groups of 10 participants each to 1) morning (am) HTN medication dosing, 2) BBTI with am HTN medication dosing, 3) nighttime non-diuretic HTN medication dosing (chronotherapy) for 6 weeks. At baseline and 6 weeks, participants will undergo 48-hour ambulatory BP monitoring, in-home sleep study, complete a 3-day bladder diary. This protocol will allow the investigators to accomplish following Aims:

Aim1: To assess the feasibility and effect of chronotherapy and BBTI in older adults with multiple comorbidities: HTN and nocturia Hypothesis 1: Chronotherapy and BBTI will be (a) feasible treatment options among comorbid older adults, and (b) nocturia and nighttime urine volume, and (c) nighttime systolic blood pressure (SBP) will have a greater decrease in BBTI and chronotherapy groups than usual care.

Aim 2: Assess safety and treatment compliance with chronotherapy. Hypothesis 2: The investigators will assess treatment compliance and also collect data on nocturnal lightheadedness and falls to begin to address the safety of HTN chronotherapy.

ELIGIBILITY:
Inclusion Criteria:

The study shall include: ambulatory and functionally-independent community-dwelling men and women aged 65+ years, with

1. nocturia ≥2/night, and
2. history of high blood pressure and receives one or more non-diuretic, once daily antihypertensive- angiotensin converting enzyme inhibitor (ACE-I), angiotensin receptor blocker (ARB), calcium channel blocker (CCB), beta blocker

Exclusion Criteria:

1. Unstable or acute medical or central nervous system conditions
2. Untreated, current, severe psychiatric condition
3. Untreated, current, severe overactive bladder syndrome
4. Post void residual > 30ml
5. Montreal cognitive assessment (MOCA) <26
6. Currently diagnosed and/or treated Obstructive Sleep Apnea, Restless Legs Syndrome, parasomnia
7. Congestive heart failure, by exam
8. Chronic kidney disease, stage III-V (eGFR<60)
9. >14 alcohol drinks per week
10. >3 caffeinated drinks (~300mg) per day

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shachi Tyagi, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started June 2022 through September 2023. The initial screening was completed telephonically and once screened eligible, the interested participants underwent study related assessments and procedures at the study research suite - Continence Research Unit at University of Pittsburgh Medical Center, Montefiore Hospital located in Pittsburgh, Pennsylvania
Pre-assignment Details: After the telephone screening, eligible participants were scheduled for the first in-person study visit. No study procedures were performed till informed consent was obtained.
Groups:
- AM (Morning) Antihypertensive Dosing- Control Arm: participants will be asked to continue taking their antihypertensive medication within an hour of awakening
  AM antihypertensive dosing: participants will be asked to continue taking their antihypertensive medication within an hour of awakening
- BBTI Arm: participants will receive the brief behavioral treatment for insomnia (BBTI) by the study nurse. Participants will also be asked to take their antihypertensive medication within an hour of awakening
  BBTI: Participants randomized to BBTI will receive 45- to 60-minute individual intervention session followed by a 30-minute follow-up session 2 weeks later, and 20-minute telephone calls after 1 and 3 weeks. BBTI will focus on four behaviors that promote sleep and discussion of homeostatic and circadian mechanisms of human sleep regulation. These four interventions are simple to conceptualize and implement, and constitute the core of efficacious multi-modal behavioral treatments for insomnia.
Period: Overall Study
Arm/Group | AM (Morning) Antihypertensive Dosing- Control Arm | BBTI Arm | PM (Evening) Antihypertensive Dosing or Chronotherapy Arm
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall, 30 participants were enrolled, 10 randomized to each of the three study arms
Groups:
- AM Antihypertensive Dosing Arm: participants will be asked to continue taking their antihypertensive medication within an hour of awakening
  AM antihypertensive dosing: participants will be asked to continue taking their antihypertensive medication within an hour of awakening
- BBTI Arm: participants will receive the behavioral treatment for insomnia BBTI by the study RN. Participants will also be asked to take their antihypertensive medication within an hour of awakening
  BBTI: Participants randomized to BBTI will receive 45- to 60-minute individual intervention session followed by a 30-minute follow-up session 2 weeks later, and 20-minute telephone calls after 1 and 3 weeks. BBTI will focus on four behaviors that promote sleep and discussion of homeostatic and circadian mechanisms of human sleep regulation. These four interventions are simple to conceptualize and implement, and constitute the core of efficacious multi-modal behavioral treatments for insomnia.
- PM Antihypertensive Dosing or Chronotherapy Arm: participants will be asked to switch their conventional once daily non-diuretic antihypertensive to bedtime
  PM antihypertensive dosing or Chronotherapy: participants will be asked to switch their conventional once daily non-diuretic antihypertensive to bedtime
- Total: Total of all reporting groups
Arm/Group | AM Antihypertensive Dosing Arm | BBTI Arm | PM Antihypertensive Dosing or Chronotherapy Arm | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (5) | 69.4 (4.6) | 71.5 (4.2) | 71.6 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 6 | 17
  Male | 6 | 3 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 9 | 7 | 10 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Participants enrolled lived in or near the city of Pittsburgh, PA
  participants
    United States | 10 | 10 | 10 | 30
Office systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 144.9 (13.3) | 137.4 (9.5) | 155.5 (14.6) | 145.8 (12.5)
Office diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 80.4 (8.3) | 79.9 (11) | 85.7 (11.7) | 82 (10.5)
Office heart rate [Mean (Standard Deviation); unit: beats per minute] | 66.5 (13.4) | 63.6 (8.7) | 68.5 (8.9) | 66.2 (10.4)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 31.2 (2.8) | 34 (8.7) | 31.4 (6.5) | 32.2 (6.4)
Post void residual [Mean (Standard Deviation); unit: ml] | 47 (75.3) | 15.7 (11.4) | 18.7 (35) | 35.4 (63.1)
Calcium channel blocker [Count of Participants; unit: Participants] | 6 | 3 | 4 | 13
Beta-blocker [Count of Participants; unit: Participants] | 3 | 5 | 1 | 9
Angiotensin converting enzyme inhibitor/ Angiotensin receptor blocker [Count of Participants; unit: Participants] | 8 | 9 | 7 | 24
Thiazide diuretic [Count of Participants; unit: Participants] | 2 | 3 | 5 | 10
Loop diuretic [Count of Participants; unit: Participants] | 1 | 1 | 0 | 2
Alpha- blocker [Count of Participants; unit: Participants] | 2 | 1 | 1 | 4
Statin [Count of Participants; unit: Participants] | 9 | 4 | 6 | 19
Antidepressant [Count of Participants; unit: Participants] | 1 | 4 | 3 | 8
Nonsteroidal anti-inflammatory drugs (NSAIDs) [Count of Participants; unit: Participants] | 0 | 0 | 2 | 2
Antimuscarinic [Count of Participants; unit: Participants] | 0 | 1 | 0 | 1
oral hypoglycemic [Count of Participants; unit: Participants] | 3 | 5 | 3 | 11
Insulin [Count of Participants; unit: Participants] | 0 | 1 | 0 | 1
Hypnotic [Count of Participants; unit: Participants] | 0 | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sleep Time Systolic Blood Pressure Dip Pre- vs Post-intervention
Description: The mean sleep time systolic blood pressure dip will be quantified by calculating the difference between daytime mean systolic pressure and nighttime mean systolic pressure expressed as a percentage of the day value for each participant across the 48-hour recording period comparing baseline and post-intervention
Time Frame: Baseline and at 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of daytime mean SBP
Arm/Group | AM Antihypertensive Dosing Arm | BBTI Arm | PM Antihypertensive Dosing or Chronotherapy Arm
Number analyzed (Participants) | 10 | 10 | 10
percentage of daytime mean SBP | -0.4 (7.9) | 7.3 (13.5) | 3.9 (10.0)
Statistical Analysis 1: Comparison: AM Antihypertensive Dosing Arm vs BBTI Arm vs PM Antihypertensive Dosing or Chronotherapy Arm; Test type: Other — Three-group ANCOVA comparisons were completed using pre- to post-intervention changes in sleep time dip in systolic BP. Analysis was adjusted for baseline value of the outcome; p = 0.65, ANCOVA

2. Secondary Outcome: Change in Nocturia Frequency Pre- vs Post-intervention
Description: change in nocturia frequency pre- vs post-intervention as determined by 3-day bladder diary completed at both time points
Time Frame: Baseline and at 6 weeks
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | AM Antihypertensive Dosing Arm | BBTI Arm | PM Antihypertensive Dosing or Chronotherapy Arm
Number analyzed (Participants) | 10 | 10 | 10
number of episodes | -0.3 (1.0) | -0.6 (0.7) | -0.3 (0.8)
Statistical Analysis 1: Comparison: AM Antihypertensive Dosing Arm vs BBTI Arm vs PM Antihypertensive Dosing or Chronotherapy Arm; Test type: Other — Three-group ANCOVA comparisons were completed using pre- to post-intervention changes in nocturia frequency. Analysis was adjusted for baseline value of the outcome; p = 0.66, ANCOVA

3. Secondary Outcome: Change in Nocturnal Polyuira Index (NPi) Pre vs Post-intervention
Description: NPi is calculated using nighttime and daytime urine volumes as reported in 3-day bladder diary as follows: NPi=(nocturnal urine volume/24-hour volume)*100
Time Frame: Baseline and at 6 weeks
Measure: Mean (Standard Deviation); unit: % of 24h urine output excreted at night
Arm/Group | AM Antihypertensive Dosing Arm | BBTI Arm | PM Antihypertensive Dosing or Chronotherapy Arm
Number analyzed (Participants) | 10 | 10 | 10
% of 24h urine output excreted at night | 0.5 (7.4) | -6.0 (9.7) | -0.9 (7.6)
Statistical Analysis 1: Comparison: AM Antihypertensive Dosing Arm vs BBTI Arm vs PM Antihypertensive Dosing or Chronotherapy Arm; Test type: Other — Three-group ANCOVA comparisons were completed using pre- to post-intervention changes in NPi. Analysis was adjusted for baseline value of the outcome; p = 0.14, ANCOVA

4. Secondary Outcome: Change in Global Pittsburgh Sleep Quality Index (PSQI) Score Pre- vs Post-intervention
Description: PSQI is a self-rated questionnaire for evaluating subjective sleep quality. PSQI global scores range from 0-21, with higher scores indicating worse sleep quality and negative change indicates sleep improvement.
Time Frame: Baseline and at 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AM Antihypertensive Dosing Arm | BBTI Arm | PM Antihypertensive Dosing or Chronotherapy Arm
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 0.5 (2.9) | -1.4 (2.2) | -1.2 (3.7)
Statistical Analysis 1: Comparison: AM Antihypertensive Dosing Arm vs BBTI Arm vs PM Antihypertensive Dosing or Chronotherapy Arm; Test type: Other — Three-group ANCOVA comparisons were completed using pre- to post-intervention changes in PSQI scores. Analysis was adjusted for baseline value of the outcome; p = 0.2, ANCOVA

5. Secondary Outcome: Change in Sleep Efficiency Pre- vs Post-intervention
Description: Sleep efficiency will be calculated as (total sleep time/time in bed)*100 with time in bed and total sleep times obtained from Zmachine worn by participants pre- and post-intervention
Time Frame: Baseline and at 6 weeks
Measure: Mean (Standard Deviation); unit: %: (total sleep time/time in bed)*100
Arm/Group | AM Antihypertensive Dosing Arm | BBTI Arm | PM Antihypertensive Dosing or Chronotherapy Arm
Number analyzed (Participants) | 10 | 10 | 10
%: (total sleep time/time in bed)*100 | -7 (15.3) | 12 (7.8) | -3 (11.8)
Statistical Analysis 1: Comparison: AM Antihypertensive Dosing Arm vs BBTI Arm vs PM Antihypertensive Dosing or Chronotherapy Arm; Test type: Other — Three-group ANCOVA comparisons were completed using pre- to post-intervention changes in sleep efficiency. Analysis was adjusted for baseline value of the outcome; p = 0.02, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of study participation for each participant, 6 weeks
Description: All participants continued to take medications that were prescribed by their outpatient providers. No dose adjustments were made either. Therefore, there was no increased risk of mortality or serious adverse events related to the study.
  We did collect adverse events were noted by self-report from participants. Specific worsening of any sleep related issues, or any falls during the study period were specifically asked during the telephonic follow-up every 2 visits following randomization.
Arm/Group | AM Antihypertensive Dosing Arm | BBTI Arm | PM Antihypertensive Dosing or Chronotherapy Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT05419830/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT05419830/ICF_001.pdf